CLINICAL TRIAL: NCT00601757
Title: Depression Intervention for Financially Disadvantaged Pregnant Women.
Brief Title: Depression Prevention for Pregnant Women on Public Assistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Caron Zlotnick, Director of Behavioral Medicine Research, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH071766 (NIH); R01MH071766 (NIH); DSIR 83-ATP
Record Dates: First submitted 2008-01-22; First posted 2008-01-28 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Depression, Postpartum; Depression
Keywords: Preventive Intervention; Postpartum Depression; Women on Public Assistance
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Participants assigned to the Postpartum Prevention Program
  Interventions: Behavioral: The Postpartum Prevention Program (PPP)
- 2 (Other): Participants assigned to enhanced care as usual
  Interventions: Behavioral: Enhanced care as usual (ECU)

INTERVENTIONS:
Behavioral: The Postpartum Prevention Program (PPP) — PPP includes interpersonal therapy sessions as well as distribution of educational material on postpartum depression. The group sessions will take place during the participant's last trimester of pregnancy. There will be four weekly sessions prior to delivery and one booster session within the first 2 weeks of the postpartum period.
  Arms: 1
Behavioral: Enhanced care as usual (ECU) — ECU includes the usual medical care provided for pregnant women at the Women's Primary Care Center at Women and Infants Hospital as well as the provision of educational material and a list of treatment resources for postpartum depression. Participants will also receive more intensive follow-up in terms of their mental health status than is typically provided in usual practice.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of an interpersonal therapy treatment called the Postpartum Prevention Program in preventing the development of postpartum depression in pregnant women who are financially disadvantaged.

DETAILED DESCRIPTION:
Postpartum depression (PPD) occurs in approximately 10% to 16% of mothers who have recently delivered babies. The impact of PPD is profound, causing considerable emotional pain for the mother as well as possible disturbances in infant development and later child adjustment. If left untreated, the mother's depression may cause strain on family life and her relationship with her child. Further research is needed to discover treatments to effectively reduce the risk of experiencing PPD. Despite preliminary findings that suggest that psychosocial treatments may prevent postpartum mood disturbances, few studies have examined the effects of preventive therapy to reduce PPD in women at risk for PPD. An area of even greater neglect is the testing of such a treatment for financially disadvantaged women, who represent a group at high risk for PPD and a group less likely to access treatment for depression than middle-class women. The Postpartum Prevention Program (PPP), an interpersonal therapy program targeting factors that may play a significant role in the development of PPD, may be helpful in reducing the occurrence of PPD. This study will compare the effectiveness of PPP to enhanced care as usual (ECU) in preventing PPD in financially disadvantaged women who are pregnant.

Participation in this single-blind study will last until 1 year after delivery. All potential participants will answer an initial questionnaire concerning stresses that may increase the risk of depression, including relationship and emotional difficulties. Selected participants will then undergo an interview about symptoms of depression, emotional difficulties, and alcohol and drug use. Participants identified as having depression will be provided appropriate referrals for treatment and their study participation will end. Participants invited to continue with the study will be randomly assigned to receive PPP or ECU. Participants assigned to receive PPP will attend four weekly 90-minute group sessions prior to delivery and one individual 50-minute booster session within 2 weeks of delivery. During these sessions, participants will learn ways to manage stress and negative feelings and how to access social support resources. Participants assigned to ECU will receive the usual medical care provided for pregnant women, educational material on PPD, and a list of referrals and resources.

All participants will complete questionnaires and interviews about their emotional difficulties, relationships with others, and use of services for these difficulties prior to treatment assignment; 4 weeks after treatment assignment; 3 weeks after delivery; and 3, 6, and 12 months after delivery. Participants will also be seen briefly at the hospital at the time of delivery and 3, 6, and 12 months after delivery to assess mother-infant relationships. All questionnaires and assessments will take between 60 and 90 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and comprehends English sufficiently to complete the study procedures
* Willing and able to receive public assistance
* Between 20 and 34 weeks of gestation
* Score of greater than 27 on the Cooper Risk Survey to identify risk of PPD

Exclusion Criteria:

* Currently receiving mental health services from a healthcare provider
* Meets criteria for a current affective disorder, anxiety disorder (excluding simple phobia), substance use disorder, or psychosis, as determined by the relevant modules of the Structured Clinical Interview for DSM-IV Nonpatient Version (SCID-NP)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2006-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Longitudinal Interval Follow-up Examination (LIFE) | Measured at Months 3, 6, and 12 postpartum

SECONDARY OUTCOMES:
Adjustment disorder or depression not otherwise specified (NOS) as measured by the Structured Clinical Interview for DSM Disorders (SCID) | Measured within Month 6 postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Caron Zlotnick, PhD, Principal Investigator — Women and Infants Hospital
Locations (3):
- United States (3):
  - Womens' Care Inc., Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Thundermist Health Center, Woonsocket, Rhode Island

REFERENCES:
- [Derived] Zlotnick C, Tzilos G, Miller I, Seifer R, Stout R. Randomized controlled trial to prevent postpartum depression in mothers on public assistance. J Affect Disord. 2016 Jan 1;189:263-8. doi: 10.1016/j.jad.2015.09.059. Epub 2015 Sep 30. PMID 26454186